CLINICAL TRIAL: NCT02579733
Title: Azathioprine Based on Endoscopy After Clinical Remission in Moderate to Severe Ulcerative Colitis
Acronym: ACE
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Not enough number of enrolling patient
Sponsor: Kyungpook National University Hospital (Other)
Collaborators: Celltrion (Industry)
Responsible Party: Principal Investigator, Eun Soo Kim, MD, PhD, Professor, Kyungpook National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: KMU-151016
Record Dates: First submitted 2015-10-16; First posted 2015-10-20 (Estimated); Last update posted 2019-08-14 (Actual); Status verified 2019-08

CONDITIONS: Ulcerative Colitis
MeSH Terms: conditions — Colitis, Ulcerative | interventions — Azathioprine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Azathioprine (Active Comparator): Azathioprine (1.5mg/kg) po for 1 year
  Interventions: Drug: Azathioprine
- Sugar pill (Placebo Comparator): Placebo drug identical to azathioprine (1.5mg/kg) po for 1 year
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Azathioprine
  Arms: Azathioprine
Drug: Placebo
  Arms: Sugar pill

SUMMARY:
The aim of this study is to determine whether azathioprine is effective for mucosal healing in UC patients who achieved clinical remission by the first course of corticosteroids but not mucosal healing in endoscopy.

DETAILED DESCRIPTION:
The sample size was calculated based on the previous study showing the difference of mucosal healing rate between azathioprine (58%) and 5-aminosalicylate (21%). With a two-tailed test of α = 0.05 and 1 - ß = 0.8, 52 patients were required.

The placebo drug which is identical to azathioprine will be provided by Celltrion drug company.

Differences in the categorical variables between the groups are examined with χ2 or the Fisher exact test. For comparisons of continuous variables, a Student t test is used.

ELIGIBILITY:
Inclusion Criteria:

* Ulcerative colitis patients with moderate to severe activity who achieved a clinical remission by the first course of corticosteroids
* Newly diagnosed or without steroid use during last 1 year
* Endoscopic Mayo subscore >0

Exclusion Criteria:

* Patients with azathioprine or biologics therapy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2016-02-01; Primary Completion 2018-12-01 (Actual); Study Completion 2018-12-01 (Actual)

PRIMARY OUTCOMES:
Mucosal healing status | one year
  Mucosal healing status will be assessed by sigmoidoscopy using Mayo endoscopic score.

CONTACTS AND LOCATIONS:
Overall Officials: Eun Soo Kim, MD, PhD, Principal Investigator — Kyungpook National University Hospital
Locations (1):
- Kyungpook National University Hospital, Daegu, South Korea

REFERENCES:
- [Derived] Hasskamp J, Meinhardt C, Patton PH, Timmer A. Azathioprine and 6-mercaptopurine for maintenance of remission in ulcerative colitis. Cochrane Database Syst Rev. 2025 Feb 27;2(2):CD000478. doi: 10.1002/14651858.CD000478.pub5. PMID 40013523